CLINICAL TRIAL: NCT01076725
Title: Insertion of the ProSeal Laryngeal Mask Airway is More Successful With the 90 Degree Rotation Technique in Pediatric Patients: a Randomized Controlled Trial
Brief Title: Rotation Technique for the Insertion of the ProSeal Laryngeal Mask Airway in Pediatric Patients
Acronym: PLMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SeoulNUBH
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2009-04

CONDITIONS: Intubation
Keywords: ProSeal LMA; standard insertion; rotational insertion

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard technique group (Active Comparator): In the standard technique group(n = 63), the PLMA was inserted by index finger insertion technique.
  Interventions: Device: Standard technique group
- Rotation technique group (Experimental): The entire cuff of the PLMA was placed in the mouth without finger insertion in a midline approach and was rotated 90 degrees counterclockwise around the tongue. The PLMA was then advanced and rotated back until resistance was felt.
  Interventions: Device: Rotation technique group

INTERVENTIONS:
Device: Standard technique group — In the standard technique group (n = 63), the PLMA was inserted by index finger insertion technique.
  Other Names: Digital insertion group
  Arms: Standard technique group
Device: Rotation technique group — The entire cuff of the PLMA was placed in the mouth without finger insertion in a midline approach and was rotated 90 degrees counterclockwise around the tongue. The PLMA was then advanced and rotated back until resistance was felt.
  Other Names: 90 degree rotation insertion
  Arms: Rotation technique group

SUMMARY:
Insertion of the ProSeal laryngeal mask airway in pediatric patients using the 90 degree rotational technique is more successful and causes less pharyngeal trauma than the standard technique in pediatric patients.

DETAILED DESCRIPTION:
In our previous series of studies, we introduced a new, simple and effective 90 degree rotational insertion technique and the insertion success rate was great and less pain occurred with the rotational technique in adult. In this study, we investigated whether the 90 degree rotational technique will improve the insertion success rate than the standard technique in pediatric patients.

We hypothesized that the 90 degree rotational technique will improve the insertion success rate and decrease the complication of 2 to 3 size PLMA than the standard index finger insertion technique in children.

One hundred twenty six Asian pediatric patients were randomly allocated to a standard technique group or rotation technique group. The size of the PLMA was from 2 to 3 according to body weight of children. In the standard technique group (n = 63), the PLMA was inserted by index finger insertion technique. In the rotation technique group (n = 63), the entire cuff of the PLMA was placed in the mouth without finger insertion in a midline approach and was rotated 90 degrees counterclockwise around the tongue. The PLMA was then advanced and rotated back until resistance was felt.

The primary outcome was success at first insertion. Secondary outcome measures were insertion time and complications.

Success at first insertion was significantly higher for the rotation technique than the standard technique, and significantly less time was required. With the rotation technique, the incidence of PLMA repositioning and blood staining was significantly less than for the standard technique.

The rotational insertion technique for PLMA is more successful than the standard insertion technique and is associated with fewer blood staining on the PLMA which suggests that it causes less pharyngeal trauma in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Asian pediatric patients (age range 3-9 years; American Society of Anesthesiologists physical status I-II) who required general anesthesia with a PLMA for elective surgery.

Exclusion Criteria:

* Pediatric patient weighed less than 10 kg or over 50 kg, had congenital heart disease, respiratory disease or were at risk of aspiration.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Insertion success rate at first attempt | 5 minute
  % of success at first trial

SECONDARY OUTCOMES:
Insertion time, sealing pressure and complication | 5 min-4 hrs
  Insertion time is an indices of the ease of insertion. Sealing pressure is an equilibrium airway pressure (maximum allowed = 40 cmH2O) when the expiratory valve of the breathing circuit was closed and a gas flow rate of 3 l/min was maintained. Blood on the surface of the cuff, incidence of postoperative sore throat or hoarseness are indices of complications.

CONTACTS AND LOCATIONS:
Overall Officials: Mija Yun, Professor, Principal Investigator — Seoul National University Bundang Hospital

REFERENCES:
- [Background] Hwang JW, Park HP, Lim YJ, Do SH, Lee SC, Jeon YT. Comparison of two insertion techniques of ProSeal laryngeal mask airway: standard versus 90-degree rotation. Anesthesiology. 2009 Apr;110(4):905-7. doi: 10.1097/ALN.0b013e31819b5d40. PMID 19293690
- [Background] Jeon YT, Na HS, Park SH, Oh AY, Park HP, Yun MJ, Kim JH, Hwang JW. Insertion of the ProSeal laryngeal mask airway is more successful with the 90 degrees rotation technique. Can J Anaesth. 2010 Mar;57(3):211-5. doi: 10.1007/s12630-009-9241-4. Epub 2010 Jan 15. PMID 20077171
- [Derived] Yun MJ, Hwang JW, Park SH, Han SH, Park HP, Kim JH, Jeon YT, Lee SC. The 90 degrees rotation technique improves the ease of insertion of the ProSeal laryngeal mask airway in children. Can J Anaesth. 2011 Apr;58(4):379-83. doi: 10.1007/s12630-010-9452-8. Epub 2011 Jan 4. PMID 21203877